CLINICAL TRIAL: NCT05342389
Title: Prospective, Randomized, Single-center Phase II Clinical Study of Camrelizumab Combined With Apatinib Versus Apaitnib Alone in the Third-line Treatment of Metastatic Gastric Cancer
Brief Title: Camrelizumab Combined With Apatinib Versus Apatinib Alone in the Third-line Treatment of Metastatic Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-II-GC-013
Record Dates: First submitted 2022-04-16; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Gastric Adenocarcinoma; Metastatic Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): A fixed dose of Camrelizumab 200mg will be administered intravenously (without preventive medication), and each infusion lasts 45min (no less than 30min, no more than 60min), once every two weeks; During the treatment period, 250 mg of Apatinib mesylate tablets will be taken orally daily continuously, and every 2 weeks is a treatment cycle. The treatment lasts for up to 2 years or until disease progression, death or intolerable toxicity occurred.
  Interventions: Drug: Camrelizumab; Drug: Apatinib Mesylate
- Control group (Active Comparator): Apatinib mesylate tablets 500 mg will be taken orally daily continuously, every 2 weeks as a treatment cycle. Treatment lasts for up to 2 years or until disease progression, death or intolerable toxicity occurs.
  Interventions: Drug: Apatinib Mesylate

INTERVENTIONS:
Drug: Camrelizumab — a PD-1 antibody
  Other Names: SHR-1210
  Arms: Experimental group
Drug: Apatinib Mesylate — an oral tyrosine kinase inhibitor
  Other Names: Ai Tan

SUMMARY:
This is a study of Camrelizumab combined with Apatinib versus Apatinib alone in the third-line treatment of metastatic gastric cancer. Paticipants will be radomized to receive treatment of Camrelizumab combined with Apatinib or Apatinib alone. The primary study hypothesis is that the adding Camrelizumab to Apatinib can prolong the progressive-free survival of the paticipants.

DETAILED DESCRIPTION:
Camrelizumab 200mg intravenously 30 - 60 min biweekly; Apatinib mesylate 250mg or 500mg oral daily continuously; The treatment lasts for up to 2 years or until disease progression, death or intolerable toxicity occurred.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, age ≥ 18 years;
2. Patients with metastatic gastric cancer confirmed by histology or cytology;
3. Baseline blood routine and biochemical indicators meet the following criteria:

1) Hemoglobin ≥ 9.0 g/dL; 2) Absolute neutrophil count (ANC) ≥ 1,500/mm3; 3) Platelet count≥ 100,000/mm3; 4) Total bilirubin ≤ 1.5 times the upper limit of normal value (ULN); 5) Alanine aminotransferase and aspartate aminotransferase ≤ 2.5 ULN; 6) The international standardized ratio of prothrombin time is ≤ 1.5, and part of the thromboplastin time is within the normal range (the lower limit of 1.2 times normal value to the upper limit of 1.2 times normal value); 7) Creatinine ≤ 1.5 ULN; 8) Urine protein <2+ (if urine protein ≥ 2+, then 24h urine protein quantitative protein must be ≤ 1g); 4．The presence of measurable lesions in patients; evaluated by investigators according to the Efficacy Evaluation Criteria (RECIST) v1.1 of Solid Tumors; 5．Eastern Tumor Collaboration Group Behavioral Status Score (ECOG PS) of 0 or 1; 6．Life expectancy ≥ 3 months; 7．The investigator assessed that the patient was able to comply with the protocol requirements; 8．Capable to sign the informed consent document.

Exclusion Criteria:

1. Patients who have undergone systemic chemotherapy, radiation therapy, surgery, hormone therapy or immunotherapy in the 2 weeks prior to the screening;
2. Patients with a history of taking apatinib;
3. Patients with hypertension that is difficult to control despite having been treated with multiple antihypertensive drugs (systolic blood pressure ≥ 160 mmHg and diastolic blood pressure ≥ 90 mmHg);
4. Patients with acute coronary syndrome (including myocardial infarction and unstable angina) within 6 months prior to admission and a history of coronary angioplasty or stenting;
5. Patients with large pleural effusions or ascites requiring drainage;
6. According to NCI-CTCAE version 5.0, patients with ≥grade 3 active infections;
7. Patients with symptomatic brain metastases;
8. Patients with partial or complete gastrointestinal obstruction;
9. Patients with interstitial lung disease with symptoms or signs of activity;
10. Patients with allergies or hypersensitivity to therapeutic drugs, patients with autoimmune diseases, and have received allogeneic tissue/solid organ transplants;
11. Patients requiring systemic corticosteroids (excluding temporary use for trials, prophylactic administration for anaphylactic reactions or to reduce swelling associated with radiotherapy) or immunosuppressants, or patients who had received such therapy less than 14 days prior to admission to this study;
12. Patients with seizures who require medication;
13. Patients who undergo major surgery (open chest surgery or laparotomy, etc.), laparotomy biopsy, trauma within 28 days before registration. Registration can be carried out on the same day of the week preceding 4 weeks (however, if an artificial anastomosis is performed without bowel resection, it should be within 14 days prior to registration);
14. Patients with unhealed wounds, unhealed ulcers or unhealed fractures;
15. Patients with a history of allergies to any of the drugs studied, similar drugs or excipients;
16. Simultaneous reception of any other anti-tumor therapy, including anti-tumor proprietary Chinese medicines and immunochemicals;
17. Pregnant, lactating women, fertile but refusing to use contraception;
18. Other situations in which the investigators determined that they were not suitable for inclusion in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 1 year
  the interval from randomization to tumor progression or death or the last follow-up

SECONDARY OUTCOMES:
Overall Survival | 2 years
  the interval from randomization to death of any reason or the last follow-up
Objective response rate | 2 years
  the proportion of subjects who achieve a best response of complete response (CR) or partial response (PR) using the RECIST 1.1 criteria
Quality of Life assessed by EORTC QLQ-OG 25 | 2 years
  The Europe Organization for Research and Treatment of Cancer,Quality of Life Questionnaire-OG 25 can assess quality of life (HRQL) in patients with tumours of the oesophagus, oesophago-gastric junction and stomach.
Toxicity assessed by CTCAE V5.0 | 2 years
  Adverse effects recorded according to CTCAE V5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jian Xiao, PhD, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliated hosipital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No